CLINICAL TRIAL: NCT04589455
Title: Determination of Pharmacokinetics and Food-effect of CBD From a Hennep Extract in Healthy Human Volunteers
Brief Title: Pharmacokinetics of CBD From a Hennep Extract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wageningen University (Other)
Collaborators: Becanex (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL74963.081.20
Record Dates: First submitted 2020-08-06; First posted 2020-10-19 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-10

CONDITIONS: CBD Pharmacokinetics
Keywords: CBD; pharmacokinetics; hennep extract; food-effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hennep extract (Experimental): A hennep extract administered in soft gel capsules in a fasted state
  Interventions: Dietary Supplement: Hennep extract
- hennep extract + high fat meal (Experimental): A hennep extract administered in soft gel capsules in a fed state
  Interventions: Dietary Supplement: Hennep extract

INTERVENTIONS:
Dietary Supplement: Hennep extract — Hennep extract from Becanex containing 70 mg CBD

SUMMARY:
Rationale: Cannabidiol (CBD) is a non-hallucinogenic plant compound of Cannabis sativa L. and has gained attention for its potential health purposes, favorable safety profile and low abuse potential. Mainly sold as food supplements, CBD-containing preparations of different composition, concentration and quality are widely available in the Netherlands via druggist stores or via Internet. However, CBD- containing preparations do not yet have a novel food status and most EU countries are currently applying a tolerance policy for CBD present in- or derived from hemp products low in THC. Likewise, there are no approved health claims for CBD, which leads to a situation that products sold by official drugstores do not contain any indication for use. Last but not least, products are not subject to any official quality control which creates a situation that consumers are unaware of the CBD content and potential contamination of the product they purchase. Getting novel food status would an important step in better regulation. Such a procedure requires a well-documented safety assessment. As part of this assessment the pharmacokinetics of CBD need to be assessed. The aim of the present study is therefore to investigate the pharmacokinetics of CBD after single oral administration of a full-spectrum hemp extract. As fatty food is reported to increase CBD oral bioavailability, we will also study the effect of a high-fat meal.

Objective: To determine the pharmacokinetics of CBD following oral administration of a novel oil-based hemp extract containing 70 mg CBD and to study the effects of a high-fat meal on the oral bioavailability of CBD.

Study design: Single dose randomized crossover intervention study Study population: healthy human volunteers, men and women from 18 to 60 years old with a BMI from 18 to 25 kg/m2.

Intervention (if applicable): In a random order, research subjects receive a single dose of hemp extract containing 70 mg CBD in soft gel capsules, both in a fasting state and with a high-fat meal.

Main study parameters/endpoints: The plasma-time curve of CBD (quantitively) and 2 of its metabolites (semi-quantitatively) after intake of the Becanex natural hemp extract. These data will be evaluated studied applying descriptive pharmacokinetic analysis (maximum peak height (Cmax), time-to-peak (Tmax), Half-life (T1/2) and area-under-the-curve (AUC)). Relative bioavailability in the fed versus fasted state will be determined by dividing individual AUC values.

ELIGIBILITY:
Inclusion criteria:

* BMI between 18,5 and 25 kg/m2
* Age between 18 and 60 years
* Weight above 50 kg
* Good general health (based on general health questionnaire)
* Veins suitable for blood sampling
* Able to speak Dutch
* Pertinent willingness to abstain from using any hemp product (including recreational Cannabis) 2 weeks prior and the entire study period.

Exclusion Criteria:

* Is currently suffering from a disease
* Has had any gastrointestinal condition/disease within the 3 months prior to the intervention
* Haemoglobin (Hb) level < 8.5 mmol/L for men and < 7.5 for women
* Has used medication in the two months before and/or during the intervention. Oral contraceptives and occasional use of NSAIDs or paracetamol (<max 3 a week on average) is allowed.
* Reported weight loss or weight gain of > 2 kg in the month prior to the intervention
* Use of herbal dietary supplements (excluding vitamins and minerals) or grapefruit products, 2 weeks before the first testday and in between the testdays.
* Allergic to products that are provided as part of the standardised diet
* Following a specific diet (e.g. vegetarian, gluten free)
* (History of) drug abuse, in this case meaning >1 x per month use of recreational drugs
* Cannabis use in the 14 days preceding the first test day.
* Smoking
* Alcohol consumption of >10 standardised glasses per week.
* Recent or planned blood donation (<3 month prior to first study day or during intervention)
* Have been pregnant or breastfeeding in the last 6 months, or plan to become pregnant during the study
* (If applicable) In case of using contraceptives, not willing to delay the break between two packets of the conception pill during which a woman gets her period during the study period.
* Personnel of Wageningen University, department of Human Nutrition and Health,
* Currently participating in other research or was participating in another study within 1 month of the intervention or within 3 months if invasive procedures were used.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-01-10 (Estimated); Primary Completion 2021-03-10 (Estimated); Study Completion 2021-03-10 (Estimated)

PRIMARY OUTCOMES:
Relative bioavailability of CBD in a fed versus a fasted state | 48 hours
  Relative bioavailability will be calculated by dividing individual AUC values
Area under the curve (AUC) | 48 hours
  Area under the curve of plasma CBD concentration after intake of a hemp extract in a fed and fasted state
Maximum concentration (Cmax) | 48 hours
  Maximum concentration of plasma CBD concentration after intake of a hemp extract in a fed and fasted state
Time to peak (Tmax) | 48 hours
  Time to peak of plasma CBD concentration after intake of a hemp extract in a fed and fasted state
Half life (t1/2) | 48 hours
  Half life of plasma CBD concentration after intake of a hemp extract in a fed and fasted state

SECONDARY OUTCOMES:
Area under the curve (AUC) | 48 hours
  Area under the curve of plasma CBD concentration after intake of a hemp extract, compared between men and women
Maximum concentration (Cmax) | 48 hours
  Maximum concentration of plasma CBD concentration after intake of a hemp extract compared between men and women
Time to peak (Tmax) | 48 hours
  Time to peak of plasma CBD concentration after intake of a hemp extract compared between men and women
Half life (t1/2) | 48 hours
  Half life of plasma CBD concentration after intake of a hemp extract compared between men and women

CONTACTS AND LOCATIONS:
Overall Officials: Ringer Witkamp, PhD, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saals BADF, De Bie TH, Osmanoglou E, van de Laar T, Tuin AW, van Orten-Luiten ACB, Witkamp RF. A high-fat meal significantly impacts the bioavailability and biphasic absorption of cannabidiol (CBD) from a CBD-rich extract in men and women. Sci Rep. 2025 Jan 29;15(1):3678. doi: 10.1038/s41598-025-87621-4. PMID 39880884